CLINICAL TRIAL: NCT01784302
Title: A 3 Arm, 5 Phase Study to Determine the Effect of Divalent and Monovalent Metal Containing Antacids and Multivitamins on the Pharmacokinetics of Raltegravir in Healthy Volunteers
Brief Title: The Effect of Antacids and Multivitamins on Raltegravir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Helen Reynolds (Other)
Responsible Party: Sponsor-Investigator, Helen Reynolds, Research nurse, University of Liverpool
Organization: University of Liverpool (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4347
Record Dates: First submitted 2013-01-28; First posted 2013-02-05 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: HIV
MeSH Terms: interventions — Geritol; Sodium Bicarbonate; aluminum hydroxide, magnesium hydroxide, drug combination; Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Maalox Plus extra (Active Comparator): Subjects will receive doses of raltegravir 400 mg and maalox plus extra
  Interventions: Drug: Maalox Plus extra; Drug: Raltegravir 400 mg
- Multivitamin (Active Comparator): Subjects will receive doses of raltegravir 400 mg along with a multivitamin tablet
  Interventions: Dietary Supplement: Multivitamins; Drug: Raltegravir 400 mg
- Sodium bicarbonate (Active Comparator): Subjects will receive doses of raltegravir 400 mg along with sodium bicarbonate
  Interventions: Dietary Supplement: Sodium bicarbonate; Drug: Raltegravir 400 mg

INTERVENTIONS:
Dietary Supplement: Multivitamins
  Arms: Multivitamin
Dietary Supplement: Sodium bicarbonate
  Arms: Sodium bicarbonate
Drug: Maalox Plus extra
  Arms: Maalox Plus extra
Drug: Raltegravir 400 mg

SUMMARY:
This study seeks to address the question of whether antacids or multivitamins influence the pharmacokinetics of raltegravir when co-administered. The aim of this study is to optimise the dosing of raltegravir when co-administered with antacids or multivitamins.

ELIGIBILITY:
Inclusion Criteria:

* The ability to understand and sign a written informed consent form, prior to participation in any screening procedures and must be willing to comply with all study requirements.
* ≥ 18 years
* Male or female subjects
* A female may be eligible to enter and participate in the study if she:
* Is of non-child-bearing potential defined as ether post-menopausal (12 months of spontaneous amenorrhea and ≥ 45 years of age)or physically incapable of becoming pregnant with documented tubal ligation, hysterectomy or bilateral oophorectomy or
* Is of child-bearing potential with a negative pregnancy test at screening and agrees to use one of the following methods of contraception to avoid pregnancy
* Complete abstinence from intercourse from 2 weeks prior to administration of IP, throughout the study and for at least 4 weeks after discontinuation of all study medication
* Double barrier method (male condom/spermicide, male condom/diaphragm, diaphragm/spermicide)
* Any intrauterine device (IUD) with published data showing that the expected failure rate is < 1 % per year
* Any other method with published data showing that the expected failure rate is < 1 % per year
* Hormonal contraception plus a barrier method. Hormonal contraception alone will not be considered adequate for inclusion into or participation in this study
* Male subjects with a female partner of childbearing potential must agree to use effective contraception as above unless vasectomized
* All subjects participating in the study will be counseled on safer sexual practices including the use of effective barrier methods (e.g. male condom)

Exclusion Criteria:

* Any significant acute or chronic medical condition
* Pregnant or lactating women
* Women of childbearing age unless using non hormonal contraception
* Evidence of organ dysfunction or any clinically significant deviation from normal during screening including laboratory determinations
* Abnormal LFTs (ALT > 2.5 x ULN, bilirubin > 1.5 x ULN)
* Positive blood screen for HIV-1 and 2 antibodies
* Positive blood screen for hepatitis B or C antibodies
* Current or recent (within 3 months) gastrointestinal disease
* Clinically relevant alcohol or drug use or history of alcohol or drug use that will hinder compliance with treatment, follow up procedures or evaluation of adverse effects
* Use of proton pump inhibitors
* Exposure to any investigational drug or placebo within 4 weeks of first dose of study drug
* Consumption of grapefruit and oranges or products containing grapefruit or oranges within 1 week of first study drug and for the duration of the study
* Use of any other drugs including over-the-counter medications and herbal preparations, within 2 weeks prior to first dose of study drug
* Previous allergy to any of the constituents of the pharmaceuticals in this trial

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-04; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in raltegravir Area under the curve (AUC)0-12h | Day 1, 6, 11, 16 and 21
  The primary endpoint will be a change in raltegravir AUC0-12 h, following dosing of antacid or multivitamin

SECONDARY OUTCOMES:
Measurement of gastrointestinal pH | Day 1, 6, 11, 16 and 21
  Correlation between gastric pH and raltegravir pharmacokinetics
Number of adverse events | Day 1 up to end of study Day 27

CONTACTS AND LOCATIONS:
Overall Officials: Saye Khoo, Prof, Principal Investigator — University of Liverpool
Locations (1):
- Royal Liverpool University Hospital, Liverpool, United Kingdom